CLINICAL TRIAL: NCT05725902
Title: A Pilot Study of the Effect of Etavopivat on Cerebral Hemodynamic Response in Children With Sickle Cell Disease
Brief Title: Study of the Effect of Etavopivat on Cerebral Hemodynamic Response in Children With Sickle Cell Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FT-4202-CBF
Record Dates: First submitted 2023-01-23; First posted 2023-02-13 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-08

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Etavopivat (Experimental): Single-arm, open-label
  Interventions: Drug: Etavopivat

INTERVENTIONS:
Drug: Etavopivat — The study intervention is etavopivat (400 mg), administered orally and once daily (QD)
  Other Names: FT-4202

SUMMARY:
An open-label, single arm study in patients 12 to 21 years of age with SCD to evaluate the effects of etavopivat on cerebral and muscle hemodynamics.

DETAILED DESCRIPTION:
This study is a pilot, open-label, single-arm study to evaluate the effect of etavopivat on cerebral hemodynamics, as measured by frequency domain near-infrared spectroscopy/diffuse correlation spectroscopy (FDNIRS/DCS) in participants 12 to 21 years of age with sickle cell disease (SCD). Cerebral blood flow (CBF), oxygen ejection fraction (OEF), and cerebral metabolic rate of oxygen (CMRO2) will be assessed FDNIRS/DCS in participants prior to, periodically throughout, and after 24 weeks of treatment with etavopivat. Approximately 12 participants will be enrolled.

The duration of study treatment will be 24 weeks. The study duration for individual participants may last up to 36 to 38 weeks and includes the Screening Period (up to 4 weeks before study treatment), the 24-week treatment period, a Safety Follow-up Visit at 4 weeks (+ 7 days) after the last dose of study drug, and an End of Study (EOS) visit approximately 8 weeks (± 7 days) after the last dose of study drug. A participant is considered to have completed the study if he or she has completed all phases of the study including the last visit or the last scheduled procedure shown in the Schedule of Events.

ELIGIBILITY:
Inclusion Criteria:

* Homozygous hemoglobin SS (HbSS) or hemoglobin S/beta0 thalassemia (HbS/β0 thal)
* Hemoglobin (Hb): Hb ≤ 9.0 g/dL at baseline
* Concomitant hydroxyurea (HU) therapy is allowed if the dose has been stable for at least 3 months with no anticipated need for dose adjustments during the study and no sign of hematological toxicity

Exclusion Criteria:

* Any one of the following requiring a medical facility visit within 14 days prior to signing the informed consent form:

  * Vaso-occlusive crisis (VOC)
  * Acute chest syndrome (ACS)
  * Splenic sequestration
  * Dactylitis
* Requires chronic transfusion therapy
* Abnormal TCD in the last 12 months
* RBC transfusion within 60 days of screening
* Severe renal dysfunction at the Screening Visit or on chronic dialysis
* Hepatic dysfunction
* Clinically relevant cardiac or pulmonary disease- e.g., congenital heart defect, uncompensated heart failure, or any unstable cardiac condition, arrhythmic heart condition, pulmonary fibrosis, pulmonary hypertension
* Major surgery involving the stomach or small intestine
* Chemotherapy or radiation within the past 2 years
* History of overt clinical stroke within previous 2 years or any history of an intracranial hemorrhage
* Clinically significant bacterial, fungal, parasitic, or viral infection currently receiving or that will require therapy
* Female who is breast feeding or pregnant

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-12-08 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Effect of etavopivat on cerebral blood flow (CBF) | 24 weeks
  Change in cerebral blood flow (CBF) assessments from baseline will be summarized with descriptive statistics by nominal study visit.
Effect of etavopivat on oxygen ejection fraction (OEF) | 24 weeks
  Change in OEF assessments from baseline will be summarized with descriptive statistics by nominal study visit.
Effect of etavopivat on cerebral metabolic rate of oxygen (CMRO2) | 24 weeks
  Change in CMRO2 assessments from baseline will be summarized with descriptive statistics by nominal study visit.

SECONDARY OUTCOMES:
Relationship between CBF and change in Hb levels | 24 weeks
  The change from baseline of CBF will be correlated to the corresponding post-baseline assessment for change in Hb.
Relationship between oxygen ejection fraction (OEF) and change in Hb levels | 24 weeks
  The change from baseline of OEF will be correlated to the corresponding post-baseline assessment for change in Hb.
Relationship between cerebral metabolic rate of oxygen (CMRO2) and change in Hb levels | 24 weeks
  The change from baseline of CMRO2 will be correlated to the corresponding post-baseline assessment for change in Hb.
Adverse events in participants with SCD | 24 weeks
  Maximum intensity of treatment emergent adverse events (TEAEs) will be summarized by system organ class and preferred term. The tabulation of deaths, serious TEAEs, serious drug-related TEAEs and TEAEs leading to study drug discontinuation will also be provided
Muscle hemodynamic effect of etavopivat on muscle blood flow | 24 weeks
  Change in muscle blood flow assessments from baseline will be summarized with descriptive statistics by nominal study visit.
Muscle hemodynamic effect of etavopivat on oxygen ejection fraction (OEF) | 24 weeks
  Change in OEF from baseline will be summarized with descriptive statistics by nominal study visit.
Muscle hemodynamic effect of etavopivat on cerebral metabolic rate of oxygen (CMRO2) | 24 weeks
  Change in CMRO2 from baseline will be summarized with descriptive statistics by nominal study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S; Amy Tang, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Emory University Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No